CLINICAL TRIAL: NCT07247682
Title: Dose-escalation of Rectal Indomethacin for Post-ERCP Pancreatitis Prevention in High-risk Patients: Protocol of a Multicentre Randomised Clinical Trial
Brief Title: Dose-escalation of Rectal Indomethacin for Preventing PEP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FirstHAnhuiMU1
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Post-ERCP Pancreatitis
Keywords: post-ERCP pancreatitis; indometacin; ERCP
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: For enhanced objectivity in data analysis, the project statisticians will be blinded to the arm allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard-dose group (Active Comparator): administration of 100 mg rectal indometacin immediately after ERCP
  Interventions: Drug: standard-dose group VS high-dose group
- high-dose group (Experimental): administration of 200 mg rectal indometacin immediately after ERCP
  Interventions: Drug: standard-dose group VS high-dose group

INTERVENTIONS:
Drug: standard-dose group VS high-dose group — A total of 1,036 eligible patients will be randomly assigned in a 1:1 ratio to one of two groups: (1) administration of 100 mg rectal indometacin immediately after ERCP (standard-dose group), or (2) administration of 200 mg rectal indometacin immediately after ERCP (high-dose group)

SUMMARY:
Our aim is to compare the efficacy of 100 mg versus 200 mg rectal indometacin in preventing post-ERCP pancreatitis (PEP) among high-risk patients without no pancreatic stenting. The 100 mg versus 200 mg indometacin trial is a multicentre, single-blind, randomized controlled study. High-risk patients for PEP without pancreatic stent insertion will be informed about the opportunity to participate. A total of 1,036 eligible patients will be randomly assigned in a 1:1 ratio to one of two groups: (1) administration of 100 mg rectal indometacin immediately after ERCP (standard-dose group), or (2) administration of 200 mg rectal indometacin immediately after ERCP (high-dose group). The primary outcome is the incidence and severity of PEP. Secondary outcomes include hyperamylasemia and other ERCP-related adverse events (AEs).

DETAILED DESCRIPTION:
Evidence suggests that escalating the rectal indometacin dose to 200 mg offers no clear advantage over the standard 100 mg regimen in high-risk patients. However, the majority of participants (76%) had received pancreatic stent placement, raising the possibility that the benefit of the supplementary strategy may have been obscured by the considerable efficacy of pancreatic stenting. Our aim is to compare the efficacy of 100 mg versus 200 mg rectal indometacin in preventing post-ERCP pancreatitis (PEP) among high-risk patients without no pancreatic stenting.

ELIGIBILITY:
Inclusion Criteria:Participants will be eligible for enrollment if they meet all of the following criteria: 1. age over 18 years; 2. classified as high risk for post-ERCP pancreatitis; 3. provision of signed, written informed consent.

Exclusion Criteria:Participants will be excluded if they meet any of the following conditions: 1. inaccessible major papilla; 2. surgically altered gastrointestinal anatomy; 3. current diagnosis of acute pancreatitis; 4. placement of a pancreatic stent; 5. contraindications to nonsteroidal anti-inflammatory drugs (NSAIDs), including known allergy, renal insufficiency, or active peptic ulcer disease; 6. anticipated low risk of post-ERCP pancreatitis (e.g., patients with chronic calcific pancreatitis, pancreatic head mass, or those undergoing biliary interventions through a pre-existing sphincterotomy); 7.severe active cardiopulmonary disease; 8. pregnancy or breastfeeding; 9. presence of an ampullary tumor.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1036 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
the incidence and severity of PEP | up to 1 months
  Patients were identified as post-ERCPpancreatitis if meeting two out of three criteria: pain consistent with acute pancreatitis; amylase or lipase>3 times normal limit; characteristic findings on imaging, in according to the Revised Atlanta International consensus.

CONTACTS AND LOCATIONS:
Overall Officials: Shaofei Wang, Principal Investigator — Department of Gastroenterology, The First Affiliated Hospital of Anhui Medical University
Locations (1):
- Department of Gastroenterology, The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
We are committed to promoting transparency and open science. Upon reasonable request and under certain conditions, individual participant data (IPD) from our study may be shared for further research. Access to the IPD will be considered on a case-by-case basis, following review and approval of a formal proposal by Qiao Mei.
  To inquire about accessing the IPD, interested parties may contact Qiao Mei at meiqiaomq@aliyun.com.
  Please note that data sharing is contingent upon meeting the criteria for ethical use, privacy, and confidentiality as outlined in our data sharing policy. Additionally, appropriate data transfer agreements may need to be established prior to sharing.